CLINICAL TRIAL: NCT07215117
Title: Engineering Whole Health Into Hospital Care to Improve Wellness: The Inpatient Whole Health Bundle
Brief Title: Engineering Whole Health Into Hospital Care - University of Michigan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sanjay Saint, Professor of Internal Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00270511; 1R18HS028963-01 (AHRQ)
Record Dates: First submitted 2025-10-08; First posted 2025-10-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Whole Health
Keywords: Holistic Health; Hospitalization; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: quasi-experimental pre-test/post-test design Note: 150 participants will give their consent for a post implementation survey. 150 participants will send their survey response in thus implying their consent to participate in the research survey. This equals 300 anticipated participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention Participants (No Intervention): Randomly selected patients who had been discharged within the 1-2 months prior to the intervention will be recruited to provide information via a survey.
- Whole Health Intervention Participants (Experimental): Hospitalized patients on the intervention units will be offered participation in the Inpatient Whole Health Bundle.
  Interventions: Behavioral: Inpatient Whole Health Bundle

INTERVENTIONS:
Behavioral: Inpatient Whole Health Bundle — Hospitalized patients on the intervention units will be offered participation in the Inpatient Whole Health Bundle, which is comprised of a variety of offerings aimed at improving the wellbeing of the patient. They can choose to use any or none of the bundle elements.
  Arms: Whole Health Intervention Participants

SUMMARY:
The purpose of this study is to test an intervention focused on improving patients' wellness and satisfaction with their hospital stay. As part of this study, patients hospitalized on specific hospital units will be asked to participate in the study intervention. This will help the researchers learn if the items offered will help improve patients' satisfaction with their hospital stay.

DETAILED DESCRIPTION:
Whole Health is a model designed to address multiple patient needs. This includes physical and spiritual wellness, personal surroundings, nutrition, relationships, and mental wellness. The Whole Health approach focuses on improving overall patient wellness and includes increased availability of complementary and alternative medicine services. While some Whole Health work is being done at outpatient facilities, this study seeks to expand and test this approach to the inpatient setting, given the potential Whole Health has for addressing patient wellness.

The goal of this study is to implement and evaluate an inpatient Whole Health Bundle intervention to improve hospitalized patients' well-being. This study will assess if implementing an Inpatient Whole Health Bundle is associated with improved patient-centric outcomes (such as perceptions of the healing environment and patient satisfaction) among hospitalized patients.

This is a quasi-experimental pre-test/post-test trial. The study will be conducted at one medical unit at the University of Michigan hospital. Study subjects will be hospitalized patients. The study will be conducted in 2 phases- pre-intervention and intervention. Each study phase will last 1-2-months. During the pre-intervention phase, a sample of patients recently discharged from the hospital will be mailed a study survey. The survey will ask questions about their satisfaction with their hospital stay.

During the intervention phase, patients staying in the hospital will be asked if they would like to participate in the study. Participants will be offered a menu of items and services that could help improve their overall well-being and their hospital stay. Patient will be free to choose or decline any of the items on the menu. A researcher will record which items, if any, a patient selects. Patients in the intervention will be mailed the same study survey as the pre- intervention phase after they are discharged from the hospital. Researchers will compare patient satisfaction responses between patients staying in the hospital during the pre- intervention phase to those who participated in the intervention. A few patients will be asked to participate in a study interview. The interviews are to better understand intervention experiences as well as barriers and facilitators to improving patient satisfaction with their hospital stay. In addition, unit level metrics will be assessed between the pre-intervention and intervention time periods.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients on medical and medical/surgical units at the University of Michigan Health System

Exclusion Criteria:

* patients that cannot speak English
* patients that are cognitively impaired or unable to provide their own consent
* patients that are under respiratory contact precautions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Whole Health Bundle and Components | 1-2 weeks post discharge
  A survey will be sent to selected patients discharged from the respective implementation units during the 1-2 months prior to implementation and to all participants in the intervention during the 1-2 month implementation period. Questions will assess if patients were offered any of the Whole Health elements and their satisfaction with those offerings. Satisfaction with each element will be assessed on a 5 point Likert scale from 1 to 5, with 1 being very dissatisfied and 5 being very satisfied
General Patient Satisfaction | 1-2 weeks post discharge
  A survey will be sent to selected patients discharged from the respective implementation units during the 1-2 months prior to implementation and to all participants in the intervention during the 1-2 month implementation period. Questions will assess overall patient satisfaction with their hospital stay. The primary measure of satisfaction will be scored on a scale of 0 to 10, where 0 is the worst hospital possible and 10 is the best hospital possible. Questions will also be asked about the care provided by their physicians and nurses while in the hospital and if the patient would recommend this hospital to friends and family.
Satisfaction with Physical Hospital Environment | 1-2 weeks post discharge
  A survey will be sent to selected patients discharged from the respective implementation units during the 1-2 months prior to implementation and to all participants in the intervention during the 1-2 month implementation period. Questions will ask about the patient's satisfaction with various aspects of the physical hospital environment using a scale of 1 - Very dissatisfied to 5- Very satisfied.

SECONDARY OUTCOMES:
Length of Stay | 4 months (2 months of pre-intervention data and 2 months of intervention data)
  Average length of stay prior to intervention will be compared to average length of stay during the intervention at the unit level for all patients regardless of study enrollment status.
Hospital Readmissions | 4 months (2 months of pre-intervention data and 2 months of intervention data)
  Total number of patients who stayed on a study unit prior to discharge and were readmitted to the hospital within 30 days of discharge will be compared to total number of patients who stayed on a study unit during the intervention period and were readmitted to the hospital within 30 days of discharge at the unit level for all patients regardless of study enrollment status.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Saint, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created. Members of the scientific community who would like a copy of the final data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing the principal investigator (Dr. Sanjay Saint). They should state their reason for requesting the data and their plans for analyzing the data. Data sets will be accompanied by a data dictionary for all study variables, both derived and raw data. The most cost-effective means for sharing data after a data-sharing agreement has been reached will be used. For example, data may be copied to a compact disk (CD) or digital versatile disk (DVD), be posted on a password protected and secure website, or made available through a third-party data archive service. Resources that are patentable and/or protectable under intellectual property rights will not be shared.
Supporting Information: Study Protocol, SAP
Time Frame: After the final publication from this study, for at least 6 years.
Access Criteria: De-identified data will be provided after requesters sign a Letter of Agreement (LOA) detailing the mechanisms by which the data will be kept secure. The LOA will also state that the recipient will not attempt to identify any individual in the data, will not share the data outside of their research team, and will provide information on any files to be linked to the data. The dataset will not include personal identifying information and all dates will be changed to integers to allow for calculation of time periods.